CLINICAL TRIAL: NCT03339570
Title: Orthopaedic Treatment of Proximal Humeral Fractures With Sling. Prospective , Non-randomized Open Study to Compare Two Treatments Effectiveness in the Management of Three-four Part (Neer's Classification) of Proximal Humeral Fractures
Brief Title: Orthopaedic Treatment Proximal Humeral Fractures
Status: Completed | Type: Observational
Sponsor: Mikel Aburto (Other)
Responsible Party: Sponsor-Investigator, Mikel Aburto, OS head of unit, Hospital General Universitario Gregorio Marañon
Organization: Hospital General Universitario Gregorio Marañon (Other)
Other Study IDs: SCIARPA 3/4
Record Dates: First submitted 2017-09-12; First posted 2017-11-13 (Actual); Results first posted 2021-11-16 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-10

CONDITIONS: Proximal Humeral Fracture
MeSH Terms: conditions — Shoulder Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Orthopedic treatment: This is the prospective cohort which includes 20 patients presenting three-four proximal humeral fracture who were treated non-surgically and followed prospectively during 12 months.
  Interventions: Procedure: Orthopedic treatment for a proximal humeral fracture

INTERVENTIONS:
Procedure: Orthopedic treatment for a proximal humeral fracture — Orthopedic treatment consisting in inmobilization of the arm in a sling for the first three weeks, followed by physical therapy.

SUMMARY:
Prospective non-randomized, open, unicentric observational study to compare two different treatments for Three-four parts fractures of proximal humerus (Neer's Classification) in elderly patients (over 75 years old). Both technics are: Sling inmobilization and shoulder arthroplasty.

DETAILED DESCRIPTION:
The investigators propose an observational study that aims to assess:

* Primarily, the functional results of a cohort of 20 pacients presenting fractures of 3 and 4 parts of proximal humerus (according to (Neer's Classification) that will be treated orthopedically (this is, non-surgically). This patients will be recruited in the emergency room of our center, and after being diagnosed of their fracture, will be treated with a sling for three weeks and subsequent rehabilitation treatment. Our intention is to assess the function of the injured shoulder using functional scales (ASES, DASH and Constant score, and VAS scale) at the time of three and twelve months from the date of the trauma.
* Secondly the investigators want to compare the results obtained in this cohort with the results of a historical cohort of patients operated in our center with the same type of fracture. Both types of treatment (non-surgical and shoulder prosthesis) are valid for this type of fracture, and endorsed by the scientific literature.

The investigators consider this to be an observational study since it assigns a single cohort of patients a single treatment (ie non-surgical treatment). The conservative treatment for this fractures is part of routine medical care, and the object of this study is to evaluate the effect of this intervention.

ELIGIBILITY:
Inclusion Criteria:

* 75 years or older.
* 3 or 4 parts fracture (Neer's Classification).

Exclusion Criteria:

* Comorbilities affecting to functional recovery.
* Fractures associating shoulder dislocation.
* Open fractures including neurovascular damage.
* Polytraumatized patients

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly population suffering proximal humeral fractures
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2019-06-16 (Actual); Study Completion 2020-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mikel Aburto, MD, Principal Investigator — HGU Gregorio Marañon
Locations (1):
- Servicio de Cirugía Ortopédica y Traumatología, HGU Gregorio Maranon, Madrid, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 patients who were enrolled after being diagnosed of a three-four parts proximal humeral fracture in the Emergency room at Hospital Gregorio Maranon (Madrid, Spain) between the years 2017 and 2019
Period: Overall Study
Arm/Group | Orthopedic Treatment
Started | 20
Completed | 16
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Orthopedic Treatment
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — All patients were recruited at Hospital Gregorio Maranon (Madrid, Spain)
  participants
    Spain | 16

OUTCOME MEASURES:

1. Primary Outcome: Constant Scale Evaluation at 3 Months and 12 Months From the Date of Trauma
Description: Changes in numeric values for the Constant shoulder function scale applied to 20 patients with fractures of 3 and 4 parts of proximal humerus (according to Neer's Classification) evaluated at the time of 3 months and 12 months from the date of the trauma.
  The Constant scale, also known as the ConstantMurley score, is one of the most widely used instruments to evaluate the shoulder. It was originally published in 1987 by the European Society of Shoulder and Elbow Surgeons (SECEC) as a method to compare function of the shoulder before and after a treatment. It is a system that combines the physical examination (65 points) with the subjective evaluation of the patient (35 points). The maximum score is 100 points, being from 90 to 100 excellent, from 80 to 89 good, from 70 to 79 average, and less than 70 poor.
Time Frame: 1 year
Population: We compared the difference in the mean value for the Constant scale measured at 3 and 12 months for the group of patients under study who treated non-surgically.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Orthopedic Treatment: Constant Scale Evaluation at 3 Months; Orthopedic Treatment: Constant Scale Evaluation at 12 Months: This is the prospective cohort which includes 20 patients presenting three-four proximal humeral fracture who were treated non-surgically and followed prospectively during 12 months.
  Orthopedic treatment for a proximal humeral fracture: Orthopedic treatment consisting in inmobilization of the arm in a sling for the first three weeks, followed by physical therapy.
Arm/Group | Orthopedic Treatment: Constant Scale Evaluation at 3 Months | Orthopedic Treatment: Constant Scale Evaluation at 12 Months
Number analyzed (Participants) | 16 | 16
units on a scale | 40.1 (9.6) | 51.8 (12.4)
Statistical Analysis 1: Comparison: Orthopedic Treatment: Constant Scale Evaluation at 3 Months vs Orthopedic Treatment: Constant Scale Evaluation at 12 Months; Student's t test was used if they were variables adjusted to a normal distribution, or the Mann-Whitney U test if they were non-normal variables; Test type: Superiority; p < 0.01, t-test, 2 sided; Mean Difference (Final Values) = 18.3

2. Primary Outcome: ASES Scale Evaluation
Description: Changes in numeric values for the ASES shoulder function scale applied to 20 patients with fractures of 3 and 4 parts of proximal humerus (according to Neer's Classification) evaluated at the time of 3 months and 12 months from the date of the trauma.
  ASES evaluation comprises a subjective part completed by the patient and an objective part performed by doctor. The subjective includes questions about pain, symptoms of instability, and activities of daily living.
  The final score includes two subscales:
  1. Pain subscale 0-50 ASES points.
  2. Function/disability subscale 0-50 ASES points. Total score 0-100 ASES points, being 0 = worse pain and functional loss/disability
Time Frame: 12 months
Population: We compared the difference in the mean value for the ASES scale measured at 3 and 12 months for the group of patients under study who treated non-surgically.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Orthopedic Treatment: ASES Scale Evaluation at 3 Months; Orthopedic Treatment: ASES Scale Evaluation at 12 Months: This is the prospective cohort which includes 20 patients presenting three-four proximal humeral fracture who were treated non-surgically and followed prospectively during 12 months.
  Orthopedic treatment for a proximal humeral fracture: Orthopedic treatment consisting in inmobilization of the arm in a sling for the first three weeks, followed by physical therapy.
Arm/Group | Orthopedic Treatment: ASES Scale Evaluation at 3 Months | Orthopedic Treatment: ASES Scale Evaluation at 12 Months
Number analyzed (Participants) | 16 | 16
units on a scale | 54.1 (16.5) | 72.4 (11.4)

3. Primary Outcome: DASH Scale Evaluation
Description: Changes in numeric values for the DASH scale applied to 20 patients with fractures of 3 and 4 parts of proximal humerus (according to Neer's Classification) evaluated at the time of 3 months and 12 months from the date of the trauma.
  DASH scale consists of 30 questions. In addition, there are two optional modules, each containing four questions, which are used to assess the symptoms and function of athletes, artists and other workers whose functional demands exceed those assessed by the DASH questionnaire.
  Calculating the final score is relatively complicated. To calculate the score it is necessary that at least 27 of the 30 questions have been answered. The final score is obtained by calculating the arithmetic mean of the answered questions, subtracting 1 and multiplying by 25. This calculation provides a score between 0 and 100, with the greater the disability the higher the score obtained, and considering variations with clinical significance those that exceed the 10 points.
Time Frame: 12 months
Population: We compared the difference in the mean value for the DASH scale measured at 3 and 12 months for the group of patients under study who treated non-surgically.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Orthopedic Treatment: DASH Scale Evaluation at 3 Months; Orthopedic Treatment: DASH Scale Evaluation at 12 Months: This is the prospective cohort which includes 20 patients presenting three-four proximal humeral fracture who were treated non-surgically and followed prospectively during 12 months.
  Orthopedic treatment for a proximal humeral fracture: Orthopedic treatment consisting in inmobilization of the arm in a sling for the first three weeks, followed by physical therapy.
Arm/Group | Orthopedic Treatment: DASH Scale Evaluation at 3 Months | Orthopedic Treatment: DASH Scale Evaluation at 12 Months
Number analyzed (Participants) | 16 | 16
units on a scale | 38.6 (20.6) | 23.8 (14.8)

4. Primary Outcome: VAS Scale Evaluation
Description: Changes in numeric values for the Changes in numeric values for the VAS scale applied to 20 patients with fractures of 3 and 4 parts of proximal humerus (according to Neer's Classification) evaluated at the time of 3 months and 12 months from the date of the trauma.
  VAS is defined as a one-dimensional scale for the subjective assessment of pain by the patient. It consists of a straight line (usually 10 centimeters -100 millimeters) in whose limits the most extreme degrees of pain intensity are located, considering a score of 0 points for the lowest degree or absence of pain (usually referred by the patient as "no pain") and 100 points for the highest grade (often referred to as "worst bearable" or "worst pain imaginable").
  The final score (from 0 to 100 points) is obtained by measuring the distance in millimeters between the lower end (score of 0 points) and the mark indicated by the patient along the line.
Time Frame: 12 months
Population: We compared the difference in the mean value for the VAS scale measured at 3 and 12 months for the group of patients under study who treated non-surgically.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Orthopedic Treatment:VAS Scale Evaluation at 3 Months; Orthopedic Treatment:VAS Scale Evaluation at 12 Months: This is the prospective cohort which includes 20 patients presenting three-four proximal humeral fracture who were treated non-surgically and followed prospectively during 12 months.
  Orthopedic treatment for a proximal humeral fracture: Orthopedic treatment consisting in inmobilization of the arm in a sling for the first three weeks, followed by physical therapy.
Arm/Group | Orthopedic Treatment:VAS Scale Evaluation at 3 Months | Orthopedic Treatment:VAS Scale Evaluation at 12 Months
Number analyzed (Participants) | 16 | 16
units on a scale | 3.3 (1.5) | 1.1 (2.1)

5. Secondary Outcome: Statistical Analysis of Changes in Numeric Values for the Constant Scale in the Context of a Cohort Study
Description: To compare the results of Constant scale at 12 months in the prospective cohort (non-surgical cohort) with the results already obtained in a historical cohort of 20 patients who were operated on by this same pathology in our hospital.
  The Constant scale, also known as the ConstantMurley score, is one of the most widely used instruments to evaluate the shoulder. It was originally published in 1987 by the European Society of Shoulder and Elbow Surgeons (SECEC) as a method to compare function of the shoulder before and after a treatment. It is a system that combines the physical examination (65 points) with the subjective evaluation of the patient (35 points). The maximum score is 100 points, being from 90 to 100 excellent, from 80 to 89 good, from 70 to 79 average, and less than 70 poor.
Time Frame: 12 months
Population: We compared difference in the mean value for the Constant scale at 12 months between the non-surgically group and a historical cohort, which consists of a group of 20 patients with a similar fracture who received a shoulder arthroplasty. Historical cohort is part of a previous study registered in Clinical Trials under the name FRALUX34, NCT02075476
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Surgical Cohort: Constant Scale Evaluation at 12 Months: The historical cohort consists of 20 patients who underwent surgery for this same pathology in our hospital, and who received a reverse total shoulder arthroplasty.
Arm/Group | Surgical Cohort: Constant Scale Evaluation at 12 Months | Orthopedic Treatment: Constant Scale Evaluation at 12 Months
Number analyzed (Participants) | 20 | 16
units on a scale | 70.1 (10.3) | 51.8 (12.4)

6. Secondary Outcome: Development of Osteonecrosis or Lack of Consolidation
Description: Collect possible complications derived from non-surgical treatment in the prospective cohort, such as humeral head osteonecrosis or lack of consolidation.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Orthopedic Treatment
Number analyzed (Participants) | 16
participants | 0

ADVERSE EVENTS:
Time Frame: Adverse effects were not recorded during the 12 months follow-up
Description: No adverse effects were collected, since it is a non-invasive treatment
Arm/Group | Orthopedic Treatment
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-01): https://cdn.clinicaltrials.gov/large-docs/70/NCT03339570/Prot_SAP_000.pdf